CLINICAL TRIAL: NCT04184882
Title: A Randomized, Double Blind, Placebo-Controlled Phase 1b Study With Open-Label Extension to Assess the Safety, Tolerability and Preliminary Efficacy of ASP0367 (MA-0211) in Pediatric Male Patients With Duchenne Muscular Dystrophy (DMD)
Brief Title: A Study to Assess the Safety, Tolerability and Preliminary Efficacy of ASP0367 (MA-0211) in Pediatric Male Participants With Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Operational Reasons
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0367-CL-0102
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: tolerability; ASP0367; MA-0211; safety
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP0367 group (Experimental): Participants will be dosed investigational product (IP) at the low dose for 2 weeks and then at the high dose for 10 weeks with the total duration of 12 weeks in the DB part and OLE part, respectively.
  Interventions: Drug: Bocidelpar
- Placebo to ASP0367 group (Placebo Comparator): Participants will be dosed matching placebo in the DB part. In OLE part, participants will dosed IP at the low dose for 2 weeks and then at the high dose for 10 weeks with the total duration of 12 weeks.
  Interventions: Drug: Bocidelpar; Drug: Placebo

INTERVENTIONS:
Drug: Bocidelpar — Oral
  Other Names: MA-0211, ASP0367
Drug: Placebo — Oral
  Arms: Placebo to ASP0367 group

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of ASP0367.

This study will also evaluate the pharmacokinetics, pharmacodynamics and efficacy on muscle function of ASP0367.

DETAILED DESCRIPTION:
This study is comprised of a 4-week pre-treatment screening period, 24-week treatment period and 4-week post-treatment follow-up period. The 24-week treatment period consists of a 12-week double-blind (DB) part and 12-week open-label extension (OLE) part and each part includes a 2 week Low dose Period and a 10-week High-dose Period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Duchenne muscular dystrophy (DMD) (confirmed by Central Genetic Counselor) defined as a clinical picture consistent with typical DMD and 1 of the following:

  * Dystrophin immunofluorescence and/or Western blot showing severe dystrophin deficiency consistent with the diagnosis of DMD.
  * Identifiable mutation within the DMD gene (deletion/duplication of 1 or more exons), where reading frame can be predicted as "out-of-frame"
  * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication or other) that is expected to preclude production of the functional dystrophin protein (i.e., nonsense mutation or deletion/duplication leading to a downstream stop codon).
* A male subject of reproductive potential (Tanner Stage 2 and above) must agree to do either of the following from screening throughout the study until 30 days after the last dose of the investigational product (IP):

  * Abstain from sexual intercourse, OR
  * If having heterosexual intercourse, must use a condom and their female partners who are of childbearing potential must use a highly effective contraception method.
* Subject has been on a stable regimen of corticosteroids for 6 months prior to the time of enrollment (at baseline).
* Subject has been on stable cardiac therapy for 3 months prior to the time of enrollment (at baseline), if used, which may include prophylactic angiotensin-converting enzyme inhibitors (ACE), angiotensin II receptor blocker (ARB), aldosterone receptor antagonists (e.g., spironolactone, eplerenone), and/or beta-blocker therapy or a combination therapy thereof.
* Subject is unable to complete the 10 meter run/walk in <6 seconds at screening.
* Subject has a PUL 2.0 entry item A score of 4, 5 or 6 at screening.
* Subject and subject's parent(s) or legal guardian agrees not to participate in another interventional study while participating in the present study.
* For those subjects receiving exon-skipping therapy, the subject has been on a stable dose regimen with a single commercially-available product for at least 6 months prior to randomization at baseline.
* For those subjects using metformin, the subject has been on a stable dose of metformin for 3 months prior to the time of enrollment (at baseline) and the investigator expects the subject to maintain the current metformin dose.

Exclusion Criteria:

* Subject has had an acute illness (i.e., upper respiratory or viral infection) within 4 weeks prior to study enrollment (at baseline), which precludes participation.
* Subject has a cardiac ejection fraction < 53% on echocardiogram at screening.
* Subject has a mean QT interval from triplicate electrocardiogram (ECG) using Fridericia's correction (QTcF) of > 450 msec at screening. If the mean QTcF exceeds the limits stated above, 1 additional triplicate ECG can be taken and utilized at screening.
* Subject has cardiac troponin I (cTnI) above the upper limit of normal (ULN) at screening and is assessed clinically significant.
* Subject has used coenzyme Q10 (CoQ10), idebenone, carnitine, or other mitochondrial focused supplements or drugs within 4 weeks prior to randomization at baseline. In addition, subject has used any peroxisome proliferator-activated receptors (PPAR) ligands such as fibrates and thiazolidinediones 4 weeks prior to randomization at baseline.
* Subject has a known or suspected hypersensitivity to ASP0367, or any components of the formulation used.
* Subject has inadequate renal function, as defined by serum Cystatin C > 2 x ULN at screening.
* Subject who has any of the following liver function tests elevated: gamma-glutamyl transferase [GGT] and/or total bilirubin [TBL]) > 1.5 x ULN at screening.
* Subject who has a positive test result for hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]), hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antigen/antibody at screening.
* Subject has mental conditions such as schizophrenia, bipolar disorder or major depressive disorder.
* Subject has a history of suicide attempt, suicidal behavior or has any suicidal ideation within 1 year prior to screening that meets criteria at a level of 4 or 5 by using the Columbia Suicide Severity Rating Scale (C-SSRS) or who is at significant risk to commit suicide, as assessed at screening or at baseline.
* Subject has severe behavioral or cognitive problems that preclude participation in the study.
* Subject has any condition, which makes the subject unsuitable for study participation.
* Subject is taking any other investigational therapy currently or has taken any other investigational therapy within 3 months prior to the time of enrollment (at baseline).
* Subject and parent/guardian are unwilling and unable to comply with scheduled visits, IP administration plan and study procedures.
* Subject tested positive for coronavirus (SARS-CoV-2) infection without any clinical signs or symptoms within 2 weeks prior to randomization at baseline and/or has had clinical signs and symptoms consistent with coronavirus (SARS-CoV-2) infection and fully recovered within 4 weeks prior to randomization at baseline.
* Subject whose parent(s) and/or caregiver(s) have increased risk of coronavirus (SARS-CoV-2) exposure from work history (e.g., nursing home, meat processing facility and correctional facility) or recent travel history unless the subject's parent(s) and/or caregiver(s) have been appropriately vaccinated with one of the COVID-19 vaccines.

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to Week 28
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment.
  A TEAE is defined as an AE observed after starting administration of the investigational product (IP) to 28 days after the last dose of IP for the double blind part or moving to the open-label extension part, whichever comes first.
  An IP-related TEAE is defined as any TEAE with a causal relationship of "yes" by the investigator.
Number of participants with vital sign abnormalities and/or AEs | Up to Week 28
  Number of participants with potentially clinically significant vital sign values.
Number of participants with body weight change abnormalities and/or AEs | Up to Week 28
  Number of participants with potentially clinically significant body weight.
Number of participants with electrocardiogram (ECG) abnormalities | Up to Week 28
  Number of participants with potentially clinically significant 12-ECG values.
Number of participants with echocardiography abnormalities and/or AEs | Up to Week 28
  Number of participants with potentially clinically significant echocardiography values.
Number of participants with laboratory value abnormalities and/or AEs | Up to Week 28
  Number of participants with potentially clinically significant laboratory values.
Number of participants with suicidal ideation and/or behavior as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline and up to Week 28
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 6 items for suicidal behavior (1. Actual attempt, 2. Interrupted attempt, 3. Aborted attempt, 4. Preparatory acts or behavior, 5. Suicidal Behavior 6. Completed suicide,) will be reported.
Change from baseline in digit span test | Baseline and up to Week 24
  The Digit span test is a subtest of Wechsler Intelligence Scale for children (WISC). This test comprises 3 parts on the fifth edition (WISC-V). Digit Span Forward requires the subject to repeat numbers in the same order as presented by the interviewer. Digit Span Backward requires the subject to repeat the numbers in the reverse order of that presented by the interviewer. Digit Span Sequencing requires the subject to sequentially order the numbers presented by the interviewer. Scores of this test are based on each raw score and total raw score.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP0367 in plasma: AUC from the time of dosing to the start of next dosing interval (AUCtau) | Up to Week 2
  AUCtau will be recorded from the PK plasma samples collected.
PK of ASP0367 in plasma: maximum concentration (Cmax) | Up to Week 2
  Cmax will be recorded from the PK plasma samples collected.
Pharmacodynamics (PD) of ASP0367: Percent change from baseline in peroxisome proliferator-activated receptor (PPAR) delta target genes expression levels in blood | Baseline and up to Week 4
  Whole blood cell samples will be collected to measure percent change in target gene expressions.
PD of ASP0367: Percent change from baseline in serum myostatin/follistatin ratio | Baseline and up to Week 12
  Serum samples will be collected to record myostatin.
Change from baseline in Performance of Upper Limb Module (PUL) (v2.0) assessment score | Baseline and up to Week 12
  The PUL Assessment v2.0 includes a total of 23 upper limb test items, with the first entry item A used to define the starting functional level. The remaining 22 items are subdivided into 3 major dimension levels as following; shoulder level (6 items, maximum score of 12), elbow level (9 items, maximum score of 17) and distal level dimension (7 items, maximum score of 13). Positive change in scores indicates an improvement.
Change from baseline on Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale | Baseline and up to Week 12
  PedsQL Multidimensional Fatigue Scale comprises the General Fatigue Scale (6 items), Sleep/Rest Fatigue Scale (6 items) and Cognitive Fatigue Scale (6 items). A 5-point response scale in each item is utilized (0 never a problem; 1 almost never a problem; 2 sometimes a problem; 3 often a problem; 4 almost always a problem). Negative change in scores indicates an improvement. This scale is based on the subject's age and will be assessed by both subject and parent or legal guardian.
Change from baseline in distance walked in 2 minutes assessed in meters | Baseline and up to Week 12
  The 2-minute walk test (2MWT) is a measurement of endurance that assesses walking distance over 2 minutes. Only ambulatory subjects conduct the 2MWT in this study.
Percent change from baseline in the assisted 6 minute cycling test (a6MCT) maximal attained revolutions | Baseline and up to Week 12
  The a6MCT has been developed as a submaximal endurance test for both legs (leg-cycling) and arms (arm-cranking) for children who are expected to lose their walking ability in the near future or are wheel chair dependent. Only arm-cranking will be applied to this study.
Change from baseline in the a6MCT maximal attained revolutions | Baseline and up to Week 12
  The a6MCT has been developed as a submaximal endurance test for both legs (leg-cycling) and arms (arm-cranking) for children who are expected to lose their walking ability in the near future or are wheel chair dependent. Only arm-cranking will be applied to this study.
Change from baseline in fat fraction by magnetic resonance spectroscopy (MRS) | Baseline, Week 12 and Week 24
  The fat fraction by MRS will be assessed for the vastus lateralis (VL) and soleus (SOL) muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Director, Study Director — Astellas Pharma Inc
Locations (5):
- United States (5):
  - University of California Davis Health, Sacramento, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Richmond at VCU, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14567&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/0367-CL-0102/